CLINICAL TRIAL: NCT03867487
Title: SGLT2 Inhibitors as a Novel Treatment for Pediatric Non-Alcoholic Fatty Liver Disease
Acronym: SLIDE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Justin Ryder (Other)
Responsible Party: Sponsor-Investigator, Justin Ryder, Vice Chair of Research for the Department of Surgery, Ann & Robert H Lurie Children's Hospital of Chicago
Organization: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 2023-6034
Record Dates: First submitted 2019-02-28; First posted 2019-03-08 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-Alcoholic Fatty Liver Disease; NAFLD; Pediatric NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double blind clinical trial in which the study team and the participants are blinded to whether the subject received placebo or study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study intervention (Experimental): Empagliflozin 10 mg will be taken daily
  Interventions: Drug: Empagliflozin 10 MG
- Control arm (Placebo Comparator): Placebo oral tablet will be taken daily
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Participants will take a 10 mg oral tablet of empagliflozin, an orally-active inhibitor of sodium-glucose co-transporter 2 (SGLT2)
  Other Names: Jardiance
  Arms: Study intervention
Drug: Placebo Oral Tablet — Participants will take an identical appearing oral tablet with zero active ingredient.
  Other Names: Control group
  Arms: Control arm

SUMMARY:
This study is a randomized, double-blind, placebo-controlled trial specifically designed to evaluate the preliminary feasibility, initial efficacy and safety of SGLT2 inhibitors for treating NAFLD in adolescents with obesity.

DETAILED DESCRIPTION:
The overall aim of this pilot study is to evaluate the feasibility and obtain a preliminary estimate of efficacy and safety of the SGLT2 inhibitor, empagliflozin, in adolescents with obesity (BMI-percentile ≥95th) who have MRI-confirmed NAFLD (hepatic fat fraction ≥ 5.5%) and have normal fasting glucose.

Participants will take empagliflozin, once daily, in the morning, with or without food, in addition to receiving lifestyle/behavioral counseling throughout the study.

The following data will be collected throughout the course of the study: Physical exam with tanner staging, safety and fasting labs, fasting blood draw (biomarkers), urine sample, stool sample, OGTT, CGM sensor placement and removal, MRI scan (MRS-Liver), BMI/anthropometrics, urine pregnancy test for female participants, iDXA scan (body fat and bone density), arterial stiffness and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

For clinical referral to screening visit:

1. Age: 12 to <20 years old
2. Diagnosis of Obesity: BMI-percentile >95th (using age- and sex- based Center for Disease Control definitions) or BMI ≥30 kg/m2
3. Elevated alanine aminotransferase (ALT) more than twice the upper limit of normal by gender (≥44 U/L for girls, ≥50 U/L for boys) within 3 months prior to screening (used for historic ALT value) OR diagnosis of NAFLD from ultrasound, MRI, or participants with biopsy-proven NASH within 12 moths of screening
4. History of lifestyle modification to treat obesity or NAFLD

To be obtained at screening visit:

1. Confirmation of Obesity
2. Tanner stage 2,3,4 or 5;
3. Normal fasting glucose tolerance (fasting blood glucose <100 mg/dL)
4. If Screening ALT is used as inclusion criteria [if > 2x historic ALT value (historical value obtained clinically within 12 months of screening visit), repeated after 4 weeks [unable to randomize until completed]]. If the repeat ALT is more than 50% increased or decreased over the screening ALT, a third ALT should be obtained. If a third ALT is not within 50% of the previous value, then the subject is ineligible but may be screened at a later date. If ALT is not used:

   * An ultrasound will be done to diagnose NAFLD if the diagnosis has not previously been made by ultrasound, MRI or biopsy
   * A MRI-derived HFF ≥ 5.5%
5. Willingness to adhere to lifestyle considerations throughout the study

Exclusion Criteria:

1. ALT > 250U/L at screening
2. History of significant alcohol intake or current use
3. Impaired fasting glucose (>100 mg/dL)
4. Diabetes (type 1 or 2)
5. Current or recent (<6 months prior to enrollment) use of weight loss medication(s)
6. Vitamin E supplementation
7. Previous bariatric surgery
8. Use of metformin
9. Prior use of empagliflozin
10. Lower limb infection/ulceration within 3 months of screening
11. Metal or magnetic implants, devices or objects inside of or on the body, which are not MRI compatible
12. Structural and functional urogenital abnormalities, that predispose for urogenital infections
13. Recent initiation (<3 months prior to enrollment) of anti-hypertensive or lipid medication(s)
14. Major psychiatric disorder
15. Known hypothalamic or pituitary dysfunction
16. Current pregnancy or plans to become pregnant

    * Females unwilling to be tested for pregnancy
    * Females who are sexually active and not protected by an effective method of birth control (e.g. IUD or medication or patch)
17. Tobacco use
18. Significant liver dysfunction (levels >5 times the upper limit of normal (ULN)):

    * ALT (ULN = 50 U/L)
    * AST (ULN = 48 U/L)
    * GGT (ULN = 48 U/L)
    * ALP (ULN = 115 U/L)
19. Platelets < 150,000 cells/mm3
20. Total bilirubin ≥ 1.3 mg/dL
21. INR ≥ 1.3
22. Albumin <3.2 g/dL
23. Gilbert's Syndrome
24. Any known causes of liver disease (except NAFLD and NASH)
25. Significant renal dysfunction (estimated glomerular filtration rate [eGFR] < 80 mL/min/1.73 m2),
26. Diagnosed monogenic obesity
27. History of cancer
28. Untreated thyroid disorder
29. History of decompensation events (ascites, variceal bleeding, hepatic encephalopathy, or hepatocellular carcinoma)
30. Current or recent (<6 months prior to enrollment) use of medication(s) associated with weight gain (e.g. atypical anti-psychotics).

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2027-05-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy as Measured by Change in Hepatic Fat Fraction (HFF) | Baseline to 26 weeks
  HFF is measured by MRI via 1H- magnetic resonance spectroscopy (MRS). HFF will be measured with single-voxel 1H-MRS on a 3.0 T Trio whole body MRI scanner, using the software package provided by the vendor. The MR elastography measurement will consist of a phase-contrast 2D GRE scan (TR/TE = 50/25 ms, matrix 256 x 90, GRAPPA R=3, slice thickness 7mm) with motion encoding in the z-direction, and acoustic excitation at 60 Hz. Four axial slices will be acquired, each with a single breath-hold. Manual ROIs covering the liver will be drawn on the stiffness maps (in kPa units) generated by the system software. Fibrosis staging will be determined following previously published guidelines.

SECONDARY OUTCOMES:
Change in Body Measurements: Body mass index (BMI) | Baseline to 26 weeks
  Height and weight will be measured using a calibrated, wall-mounted stadiometer and an electronic scale, respectively. Three consecutive height and weight measurements will be obtained and averaged. BMI will be calculated as the weight in kilograms divided by the height in meters, squared.
Change in Body Measurements: Body Fat % | Baseline to 26 weeks
  Total percent body fat mass and lean muscle mass will be determined by dual energy x-ray absorptiometry (iDXA, GE Healthcare). Body fat percentage is calculated by body fat mass divided by the sum of fat and lean masses.
Change in Body Measurements: Visceral Fat % | Baseline to 26 weeks
  Total body fat mass and visceral fat mass will be determined by dual energy x-ray absorptiometry (iDXA, GE Healthcare). Visceral fat percentage of total body mass is calculated by visceral fat mass divided by the sum of total fat and lean masses. Visceral fat percentage of total fat mass is calculated by visceral fat mass divided by total fat mass.
Change in Biomarkers of NAFLD: Alanine transaminase (ALT) | Baseline to 26 weeks
  Fasting (≥12 hours) blood will be collected for the measurement of ALT at Fairview Diagnostics Laboratories, Fairview-University Medical Center, Minneapolis, MN - a Center for Disease Control and Prevention certified laboratory.
Change in Biomarkers of NAFLD: Cytokeratin (CK)-18 | Baseline to 26 weeks
  Fasting plasma samples will be used to measure CK-18 via Luminex Multiplex platform (Millipore, St. Louis, MO).
Change in Blood Pressure | Baseline to 26 weeks
  Blood pressure measurements will be obtained manually on the same arm using the same cuff size and equipment. Standardized procedures will be employed as described in previously published standards. Individual cuff size will be determined by measuring the arm circumference midway between the acromial process and the bony olecranon. Sitting blood pressure and heart rate will be measured after the participant has been resting quietly without legs crossed for 10 minutes. Measurements will be made three consecutive times (3-minute intervals). The final two of three independent measurements will be averaged.
Change in Arterial Stiffness | Baseline to 26 weeks
  Carotid- and femoral artery augmentation index and carotid-femoral pulse wave velocity (PWV) will be measured by the SphygmoCor® MM3 system (AtCor Medical, Sydney, Australia). Augmentation index is a measure of the relative magnitude of the reflected (or retrograde) pulse wave early in the cardiac cycle. Higher values of augmentation index represent increased arterial stiffening. PWV will be calculated as distance divided by transit time. Since pulse wave transit time decreases in stiffer arterial segments, higher values of pulse wave velocity represent increased arterial stiffness.
Change in Glycemic Control | Baseline to 26 weeks
  After fasting measures are completed, we will perform a 2-hour oral glucose tolerance test with fasting (-15 and 0-min) and serial postprandial (15-, 30-, 45-, 60-, 90-, and 120-minutes) plasma concentrations of glucose (glucose oxidase, YSI INC., Yellow Sprigs, OH) and insulin (ELISA, ALPCO Diagnostics, Windham, NH) measured after administration of a 75g glucose challenge. Samples will be batched and a stored for analysis at the completion of the study. Insulin sensitivity will be estimated by the whole-body insulin sensitivity index (WBISI) using plasma glucose and insulin concentrations.
Change in Proton Density Fat Fraction (PDFF) from MRI | Baseline to 26 weeks
  A proton density fat fraction (PDFF) image will be acquired using LiverLab's "qdixon" imaging acquisition (3D gradient echo, TR=9ms, flip angle=4°, TE=1.15, 2.46, 3.69, 4.92, 6.15, 7.38 ms, 2x2x3.5mm resolution, one 17s breath-hold). The MRS measurement of HFF will be used as the primary metric. As a secondary endpoint we will use PDFF which has shown promise as a measure of fibrosis staging compared to liver biopsy in children.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ryder, PhD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No